CLINICAL TRIAL: NCT06412809
Title: Combined Land- and Water-Based Core and Lower Extremity Strength Training in Improving the Jump Performance Among Volleyball and Basketball Players: A Randomized Controlled Trial
Brief Title: Combined Land- and Water-Based Core and Lower Extremity Strength Training in Improving the Jump Performance Among Volleyball and Basketball Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mariano Marcos State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PT-001
Record Dates: First submitted 2024-05-08; First posted 2024-05-14 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Athletes
Keywords: Strength training; Core strengthening; Jump performance; Basketball players; Volleyball exercise

STUDY DESIGN:
Intervention Model Description: Volleyball and basketball players
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors are blinded to the grouping of the participants and the interventions of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Combined Land- and Water-Based Exercise (Experimental): Core and lower extremity strengthening exercises done on both land and water.
  Interventions: Other: Combined Land- and Water-Based Exercise
- Land-Based Exercise (Active Comparator): Core and lower extremity strengthening exercises that are implemented solely on land.
  Interventions: Other: Land-Based Exercise
- Water-Based Exercise (Active Comparator): Core and lower extremity strengthening exercises that are implemented solely in water.
  Interventions: Other: Water-Based Exercise

INTERVENTIONS:
Other: Combined Land- and Water-Based Exercise — Strengthening exercises targeting the core and lower extremities (quadriceps, hamstring, and gastrocnemius) were implemented both on land and in water. The exercises are done for approximately one hour/day, three days/week for two consecutive weeks. The following are the included exercises:
  Land-based exercise:
  1. Plank exercise
  2. Russian twist
  3. Push-up
  4. Goblet squat
  5. Kettle bell swing
  Water-based exercise:
  1. Flutter kicks
  2. Isometric core crunches
  3. Jump lunges
  4. Kicks
  5. Resisted knee flexion
  Arms: Combined Land- and Water-Based Exercise
Other: Land-Based Exercise — Strengthening exercises targeting the core and lower extremities (quadriceps, hamstring, and gastrocnemius) were implemented on land. The exercises are done for approximately one hour/day, three days/week for two consecutive weeks. The following are the included exercises:
  1. Plank exercise
  2. Russian twist
  3. Dead bug
  4. Push-up
  5. Goblet squat
  6. Nordic hamstring curl
  7. Lunges
  8. Kettle bell swing
  9. Calf raises
  10. Bird dog
  Arms: Land-Based Exercise
Other: Water-Based Exercise — Strengthening exercises targeting the core and lower extremities (quadriceps, hamstring, and gastrocnemius) were implemented in the water. The exercises are done for approximately one hour/day, three days/week for two consecutive weeks. The following are the included exercises:
  1. Core pulls
  2. Flutter kicks
  3. Water cycling
  4. Isometric core crunches
  5. Seated push-up
  6. Jump squats
  7. Jump lunges
  8. Kicks
  9. Ankle jumps
  10. Resisted knee flexion
  Arms: Water-Based Exercise

SUMMARY:
Given conflicting studies regarding the effect of land-based and water-based training on the jump performance of volleyball and basketball players, a randomized controlled trial is conducted. This study hypothesizes that combined land- and water-based core and lower strength training significantly increase jump performance of volleyball and basketball players in comparison to either land- and/or water-based training alone.

DETAILED DESCRIPTION:
Numerous studies focused on the effect of sole land- or water-based exercise training to improve either core and/or lower extremities alone, which could result in improved jump performance. With the continuously increasing popularity of volleyball and basketball, where players get better and better, competition in these fields is also heightened. Hence, identifying other methods to improve game performance, such as improving muscle strength and jump performance can be explored to contribute to the existing literature and could benefit the volleyball and basketball players themselves, trainers/coaches, universities competing in sports competitions locally, nationally, and even internationally, and to physical therapists who are venturing to sports physical therapy.

The study then seeks to investigate whether combined land- and water-based exercises targeting the core and lower extremity muscle strength can enhance the jump performance of basketball and volleyball players. With this, a three-arm, single-blinded randomized controlled trial is being conducted among basketball and volleyball players. Participants are grouped into combined land- and water-based exercise, land-based exercise, and water-based exercise.

To proceed with the implementation, the researchers acquired ethical clearance from the MMSU Ethics and Review Board. Recruitment of participants happened within a University at Ilocos Norte, Philippines. Acquisition of informed consent was done before other screening procedures to identify the eligibility of participants to participate in the study. Eligible participants were randomized accordingly to either the three (3) aforementioned groups.

The exercises implemented in each group are based on existing literature regarding their effect on either the core or lower extremity strength, and combined to create a new and applicable exercise program, These exercise programs were also verified applicable by two licensed physical therapists who are also well-versed in strength training protocols. The participants are being trained accordingly one hour/day, three days/week for two consecutive weeks.

As to the pre-and post-test measurements of the primary and secondary outcomes, assessment is done by two independent licensed physical therapists who are blinded to the participants and interventions. Moreover, the assessors are well-versed in the assessment of the different outcome measurements (Plank core strength test, 1RM, 10-meter Sprint Test, Margaria-Kalaman Power Test) and in using the MyJump Lab Mobile App, duly purchased by the researchers, used for the assessment of countermovement jump and squat jump.

The SPSS version 22 will be used for data analysis by an independent statistician. Descriptive and comparative statistics will be used to analyze all data within- and between-groups, respectively. For the descriptive statistics, frequency, percentages, mean, and standard deviation will be utilized, while the two-way ANOVA and/or the paired T-test will be utilized for the comparative statistics.

ELIGIBILITY:
Inclusion Criteria. Volleyball and basketball players, specifically who:

* are at least 18 years-old,
* are enrolled in an Ilocos-based university during the second semester of academic year 2023-2024,
* played in at least one (1) official university-wide game,
* are physically prepared for the training, which is identified using the Physical Activity Readiness Questionnare for Everyone (PAR-Q+), and
* have provided informed consent.

Exclusion Criteria: Volleyball and basketball players who:

* sustained injuries within 6 weeks before the start of the study,
* have uncontrolled angina, uncontrolled hypertension, uncontrolled dysrhythmias, recent history of congestive heart failure, and/or severe aortic valve disease,
* has condition/s that is/are contraindicated for pool therapy such as open wounds, skin infections, high fever, incontinence, fear of water, etc.,
* answered "Yes" to at least one question from the PAR-Q+; and
* declined to participate.

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2024-04-26 (Actual); Primary Completion 2024-05-12 (Actual); Study Completion 2024-05-17 (Actual)

PRIMARY OUTCOMES:
Vertical Jump | 2 weeks
  This outcome measure is assessed using the manual vertical reach test technique. Unit of measurement is in centimeters (cm). Pre- and post-test measurement will be gathered.
Countermovement Jump | 2 weeks
  This outcome measure is assessed using the MyJump Lab Application. Unit of measurement is in centimeters (cm). Pre- and post-test measurement will be gathered.
Squat Jump | 2 weeks
  This outcome measure is assessed using the MyJump Lab Application. Unit of measurement is in centimeters (cm). Pre- and post-test measurement will be gathered.

SECONDARY OUTCOMES:
Core Strength | 2 weeks
  Best time for plank will be assessed, measured in seconds (s). Pre- and post-test measurement will be gathered.
Quadriceps-Hamstring Strength | 2 weeks
  This outcome measure used the 1RM of the participant, measured in pounds (lbs), as measurement of Quadriceps-Hamstring strength. Pre- and post-test measurement will be gathered.
Gastrocnemius strength | 2 weeks
  This outcome measure will simply use the Manual Muscle Test (MMT) as the basis, using scale method as elaborated by Brown and Avers (2019)'s Manual Testing 10th edition. Pre- and post-test measurement will be gathered.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Audrey D Viloria, Study Chair — Mariano Marcos State University
Locations (1):
- Mariano Marcos State University, Batac, Il, Philippines

IPD SHARING:
Plan to Share IPD: No
Based on the approved ethical considerations of the study by the ethics review board, the raw data will be kept with utmost confidentiality for at most five years. It can be viewed if required by the public, but with limitations, such as the provision of code names of participants to abide with data privacy.

REFERENCES:
- [Background] Gabbett TJ. The development of a test of repeated-sprint ability for elite women's soccer players. J Strength Cond Res. 2010 May;24(5):1191-4. doi: 10.1519/JSC.0b013e3181d1568c. PMID 20386127
- [Background] Wirth K, Keiner M, Fuhrmann S, Nimmerichter A, Haff GG. Strength Training in Swimming. Int J Environ Res Public Health. 2022 Apr 28;19(9):5369. doi: 10.3390/ijerph19095369. PMID 35564764
- [Result] Balsalobre-Fernandez C, Glaister M, Lockey RA. The validity and reliability of an iPhone app for measuring vertical jump performance. J Sports Sci. 2015;33(15):1574-9. doi: 10.1080/02640414.2014.996184. Epub 2015 Jan 2. PMID 25555023
- [Result] Seo DI, Kim E, Fahs CA, Rossow L, Young K, Ferguson SL, Thiebaud R, Sherk VD, Loenneke JP, Kim D, Lee MK, Choi KH, Bemben DA, Bemben MG, So WY. Reliability of the one-repetition maximum test based on muscle group and gender. J Sports Sci Med. 2012 Jun 1;11(2):221-5. eCollection 2012. PMID 24149193
- [Result] Bishop C, Jarvis P, Turner A, Balsalobre-Fernandez C. Validity and Reliability of Strategy Metrics to Assess Countermovement Jump Performance using the Newly Developed My Jump Lab Smartphone Application. J Hum Kinet. 2022 Sep 8;83:185-195. doi: 10.2478/hukin-2022-0098. eCollection 2022 Aug. PMID 36157951
- [Result] Gencoglu C, Ulupinar S, Ozbay S, Turan M, Savas BC, Asan S, Ince I. Validity and reliability of "My Jump app" to assess vertical jump performance: a meta-analytic review. Sci Rep. 2023 Nov 17;13(1):20137. doi: 10.1038/s41598-023-46935-x. PMID 37978338
- [Result] Hetzler RK, Stickley CD, Lundquist KM, Kimura IF. Reliability and accuracy of handheld stopwatches compared with electronic timing in measuring sprint performance. J Strength Cond Res. 2008 Nov;22(6):1969-76. doi: 10.1519/JSC.0b013e318185f36c. PMID 18978613
- [Result] TY - JOUR AU - Selvakumar, Kiruthika AU - Manoharlal, Manoj AU - Rusli, Nadia AU - Jing, Low AU - Thirruvevenkadam, Ilayaraja PY - 2021/06/01 SP - 04 EP - 10 T1 - Effectiveness of Modified Plank vs Conventional Plank on Core Muscle Endurance and Stability in Recreational Athletes: A Quasi-Experimental study VL - 15 DO - 10.7860/JCDR/2021/48224.15043 JO - Journal of Clinical and Diagnostic Research ER -
- [Result] TY - JOUR AU - Keiner, Michael AU - Kadlubowski, Björn AU - Hartmann, Hagen AU - Stefer, Tobias AU - Wirth, Klaus PY - 2021/05/05 SP - T1 - The Influence of Maximum Strength Performance in Squats and Standing Calf Raises on Squat Jumps, Drop Jumps, and Linear as well as Change of Direction Sprint Performance in Youth Soccer Players VL - DO - 10.23937/2469-5718/1510190 JO - ER -
- [Result] Cuthbert M, Ripley N, McMahon JJ, Evans M, Haff GG, Comfort P. The Effect of Nordic Hamstring Exercise Intervention Volume on Eccentric Strength and Muscle Architecture Adaptations: A Systematic Review and Meta-analyses. Sports Med. 2020 Jan;50(1):83-99. doi: 10.1007/s40279-019-01178-7. PMID 31502142
- [Result] Jonhagen S, Ackermann P, Saartok T. Forward lunge: a training study of eccentric exercises of the lower limbs. J Strength Cond Res. 2009 May;23(3):972-8. doi: 10.1519/JSC.0b013e3181a00d98. PMID 19387378
- [Result] Collins KS, Klawitter LA, Waldera RW, Mahoney SJ, Christensen BK. Differences in Muscle Activity and Kinetics Between the Goblet Squat and Landmine Squat in Men and Women. J Strength Cond Res. 2021 Oct 1;35(10):2661-2668. doi: 10.1519/JSC.0000000000004094. PMID 34341315
- [Result] Lake JP, Lauder MA. Kettlebell swing training improves maximal and explosive strength. J Strength Cond Res. 2012 Aug;26(8):2228-33. doi: 10.1519/JSC.0b013e31825c2c9b. PMID 22580981
- [Result] Dell'Antonio E, Ruschel C, Hubert M, Lucas RD, Haupenthal A, Roesler H. The Effect of Aquatic Plyometric Training on Jump Performance Including a Four-week Follow-up in Youth Female Volleyball Players. J Hum Kinet. 2022 Sep 8;83:197-205. doi: 10.2478/hukin-2022-0058. eCollection 2022 Aug. PMID 36157943
- [Result] TY - JOUR AU - Roush, James AU - Heick, John AU - Genovese, Joseph AU - Kurashima, Kyle AU - Yarrington, Dallin PY - 2020/01/01 SP - T1 - Using Kinetic Energy with Potential Energy When Determining Power During the Stair Climbing Test VL - DO - 10.46743/1540-580X/2020.1928 JO - Internet Journal of Allied Health Sciences and Practice ER -